CLINICAL TRIAL: NCT03020407
Title: The Randomized Controlled Trial of Inferior Vena Cava Ultrasound-guided Fluid Management in Septic Shock Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 589/59
Record Dates: First submitted 2017-01-03; First posted 2017-01-13 (Estimated); Results first posted 2021-08-30 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-04

CONDITIONS: Septic Shock
Keywords: Septic Shock; Inferior vene cava diameter; Resuscitation; Mortality
MeSH Terms: conditions — Shock, Septic | interventions — Anti-Bacterial Agents; Anti-Infective Agents; Vasoconstrictor Agents; Norepinephrine; Dopamine; Epinephrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVC Ultrasound-guided (Experimental): The treating physician will promptly assess the IVC diameter to obtain the collapsibility index (IVCCI) (or distensibility index, IVCDI) of an eligible patient. A previous study showed that IVCCI > 40% were strongly associated with fluid responsiveness. Accordingly, the patient will be given 10 ml/kg of bolus of 0.9% normal saline solution (NSS) each time when the IVCCI > 40% is discovered and serial measurements will be done after each intravenous bolus is achieved until the IVCCI < 40 % during our protocol. Prompt empirical antibiotics will be given to the patients within one hour before the treatment allocation.
  Interventions: Procedure: IVC Ultrasound-guided; Drug: Antibiotics; Drug: Vasopressor
- Usual care (No Intervention): Patients will be promptly and empirically treated by 30 ml/kg loading of NSS in this treatment arm. After the NSS bolus, treatment with either the additional intravenous fluid or a vasopressor is given depended on physicians' discretion during the 6-hour study period. Prompt empirical antibiotics will be given to the patients within one hour before the treatment allocation.

INTERVENTIONS:
Procedure: IVC Ultrasound-guided — IVC is identified in longitudinal section in the subcostal area of a patient using the curvilinear probe of standard ultrasound. The selected area of IVC diameter measurement is set at 2 centimeters distal to the confluence of hepatic vein by M-mode coupled by two-dimensional mode on frozen screen images using the Sonosite® X-porte.
  Arms: IVC Ultrasound-guided
Drug: Antibiotics — Prompt empirical antibiotics will be given to the patients within one hour before the treatment allocation.
  Other Names: Antimicrobials
  Arms: IVC Ultrasound-guided
Drug: Vasopressor — The threshold to the need of a vasopressor is set at mean arterial pressure below 65 mmHg if a patient's condition does not response to the fluid therapy.
  Other Names: Norepinephrine, dopamine, epinephrine
  Arms: IVC Ultrasound-guided

SUMMARY:
The primary aim of this study is to evaluate the 30-day mortality outcome of the septic shock patients who are treated with ultrasound-assisted fluid management using change of the inferior vene cava (IVC) diameter during respiratory phases in the first 6 hours compared with those treated with "usual-care" strategy.

DETAILED DESCRIPTION:
Septic shock (SS) is globally prevalent in with high mortality rate.The current focuses on initial treatment of this condition emphasize on the early recognition, prompt administration of antibiotic, and restoration of hemodynamic with aggressive fluid resuscitation and vasopressor. Regarding the initial fluid therapy, administration of empirical crystalloid at the dose of 30 ml/kg is recommended in the guideline. The ultrasound-assisted management of shock patients has been introduced in the past decade and now is widely used. By using the measurement of inferior vena cava (IVC) diameter change during respiratory phases, physicians can predict the fluid responsiveness in the shock patients and tailor the fluid therapy during the resuscitation.Unfortunately, clinical outcome related to the use of this concept in SS resuscitation has not been well studied. Inadequate resuscitation with fluid therapy is related with higher mortality; however, fluid bolus or positive fluid balance that may result from "too aggressive" fluid administration is also associated with increased mortality in SS patients. The primary aim of this study was to evaluate the 30-day mortality outcome of the SS patients who were treated with ultrasound-assisted fluid management using change of the IVC during respiratory phases in the first 6 hours compared with those who were treated with "usual-care" strategy. The secondary outcomes were to compare the rate of the need for mechanical ventilation (MV) and renal replacement therapy (RRT) as well as the 6-hours lactate clearance and the change in Sequential Organ Failure (SOFA) score in 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patient who attended the emergency department with septic shock (defined by those who require a vasopressor to maintain a mean arterial pressure (MAP) of 65 mm Hg or greater and whose serum lactate level greater than 2 mmol/L in the absence of hypovolemia.)

Exclusion Criteria:

* 1) Congestive pulmonary edema or known to have poor systolic cardiac function (left ventricular ejection fraction ≤ 40%).
* 2) Known to have right heart pathologies.
* 3) Having or suspected to have marked ascites, significant bowel dilatation or the conditions that can cause abdominal hypertension.
* 4) Body mass index ≥ 30 kg/square meter.
* 5) Having concomitant attack of severe airway disease (eg. Asthma, COPD) that may have confounded the IVC interpretation due to the positive intrathoracic pressure.
* 6) IVC can not be identified or its diameter cannot be measured correctly.
* 7) Having end-stage renal diseases with or without dialysis.
* 8) Having non-infectious diseases as final diagnoses.
* 9) Pregnant women.
* 10) Have been referred or treated from other healthcare facility.
* 11) Having active hemorrhages.
* 12) Duplicated cases.
* 13) who had "do-not-resuscitate" living will.
* 14) Declined to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khrongwong Musikatavorn, MD, Principal Investigator — Emergency Unit, Faculty of Medicine, Chulalongkorn Hospital
Locations (1):
- Emergency Medicine Unit, King Chulalongkorn Memorial Hospital, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Musikatavorn K, Plitawanon P, Lumlertgul S, Narajeenron K, Rojanasarntikul D, Tarapan T, Saoraya J. Randomized Controlled Trial of Ultrasound-guided Fluid Resuscitation of Sepsis-Induced Hypoperfusion and Septic Shock. West J Emerg Med. 2021 Feb 10;22(2):369-378. doi: 10.5811/westjem.2020.11.48571. PMID 33856325

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IVC Ultrasound-guided | Usual Care
Started | 105 | 106
Completed | 101 | 101
Not Completed | 4 | 5
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 2 | 3
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IVC Ultrasound-guided | Usual Care | Total
Number analyzed (Participants) | 101 | 101 | 202
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 49 | 96
  >=65 years | 54 | 52 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (20.1) | 63.7 (16.8) | 64.5 (18.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 38 | 86
  Male | 53 | 63 | 116
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 101 | 101 | 202
Region of Enrollment [Count of Participants; unit: Participants]
  Thailand | 101 | 101 | 202
Patients with infections [Count of Participants; unit: Participants] | 101 | 101 | 202

OUTCOME MEASURES:

1. Primary Outcome: 30-day Mortality
Description: 30-day mortality related to septic shock
Time Frame: 30 day after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | IVC Ultrasound-guided | Usual Care
Number analyzed (Participants) | 101 | 101
Participants | 20 | 19

2. Secondary Outcome: Percentage Change of 6-hour Lactate
Description: The percentage change in blood lactate at 6 hour after initiation of treatment, calculated by [(Initial blood lactate level at presentation - blood lactate level at 6 hours after treatment)/Initial blood lactate level at presentation] x 100%. The higher positive value means the more relative reduction of blood lactate after treatment from that of initial presentation and indicates a better clinical outcome.
Time Frame: 6 hours after treatment
Population: Data of 6-hour lactate was obtained among 100 patients (missing data in one patient) in the Usual care group and 100 patients (missing data in one patient) in the IVC Ultrasound-guided group .
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | IVC Ultrasound-guided | Usual Care
Number analyzed (Participants) | 100 | 100
percentage change | 39.2 [7.4 to 60] | 35.9 [16.3 to 65.5]

3. Secondary Outcome: 6-hour Cumulative Amount of Intravenous Fluid (mL)
Description: Cumulative amount of intravenous fluid (mL) during the first 6 hours after treatment.
Time Frame: 6 hours after treatment
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | IVC Ultrasound-guided | Usual Care
Number analyzed (Participants) | 101 | 101
mL | 1900 [1500 to 2570] | 2600 [2300 to 3220]

4. Secondary Outcome: 72-hour Cumulative Amount of Intravenous Fluid (mL) After Treatment
Description: Cumulative amount of intravenous fluid (mL) during the first 72 hours after treatment.
Time Frame: 72 hours after treatment
Population: Data of 72-hour cumulative amount of intravenous fluid was available among 83 patients (missing data in 18 patients; 6 discharge within 72 hours, 5 transfer out, 4 missing records and 3 death within 72 hours) in the Usual care group and 79 patients (missing data in 22 patients, 10 discharge within 72 hours, 4 transfer out, 3 missing records, 5 death within 72 hours) in the IVC Ultrasound-guided group .
Measure: Mean (Inter-Quartile Range); unit: mL
Arm/Group | IVC Ultrasound-guided | Usual Care
Number analyzed (Participants) | 79 | 83
mL | 7,300 [5040 to 9200] | 7,702 [5900 to 11275]

5. Secondary Outcome: Change in Sequential Organ Failure Assessment (SOFA) Score in 72 Hours After Treatment
Description: The change in Sequential Organ Failure Assessment (SOFA) score between the score at initial presentation and 72 hours after treatment, determined by SOFA score at presentation minus the SOFA score at 72 hours after treatment. The possible minimum and maximum value of the change in SOFA score are -24 and +24, respectively. The higher value means the more relative reduction in SOFA score at 72 hours and indicates a better clinical outcome.
Time Frame: 72 hours after treatment
Population: Data of 72-hour cumulative amount of intravenous fluid was available among 86 patients (missing data in 15 patients; 6 discharge within 72 hours, 5 transfer out, 1 lack of sufficient information and 3 death within 72 hours) in the Usual care group and 78 patients (missing data in 23 patients, 10 discharge within 72 hours, 4 transfer out, 4 lack of sufficient information, 5 death within 72 hours ) in the IVC Ultrasound-guided group .
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | IVC Ultrasound-guided | Usual Care
Number analyzed (Participants) | 78 | 86
Score on a scale | 1 [-1 to 3] | 1 [-1 to 2]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | IVC Ultrasound-guided | Usual Care
All-Cause Mortality (participants affected / at risk) | 20/101 | 19/101
Serious Adverse Events (participants affected / at risk) | 31/101 | 35/101
Other Adverse Events (participants affected / at risk) | 4/101 | 2/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVC Ultrasound-guided (N=101) | Usual Care (N=101)
Renal replacement therapy (Renal and urinary disorders) | 8 (8) | 5 (5)
Mechanical ventilator (Respiratory, thoracic and mediastinal disorders) | 23 (23) | 30 (30)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVC Ultrasound-guided (N=101) | Usual Care (N=101)
Acute kidney injury (Renal and urinary disorders) | 4 (101) | 2 (101)

LIMITATIONS AND CAVEATS:
This study was conducted with the specific study protocol at a single, tertiary-care hospital. Second, physicians should use cautious clinical judgment or different approaches in different types of patients. The interpersonal variation and sampling position may have affected the consistency of IVC diameter measurement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT03020407/Prot_SAP_000.pdf